CLINICAL TRIAL: NCT00413790
Title: A 3-Way Cross-Over, Randomized, Placebo-Controlled, Double-Blind, Multicenter Study to Assess the Pharmacologic Effects of a 7-Day Exposure to Darifenacin 15 mg o.d. and Tolterodine ER 4 mg o.d on Cardiovascular Parameters in Healthy Subjects 50 Years of Age and Older
Brief Title: Pharmacologic Effects of Darifenacin and Tolterodine on Cardiovascular Parameters in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Procter and Gamble (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CDAR328A2413
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Healthy
Keywords: Heart rate, overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — darifenacin; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): Darifenacin
  Interventions: Drug: Darifenacin
- 2 (Active Comparator): Tolterodine
  Interventions: Drug: Tolterodine
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darifenacin — Darifenacin tablets 15 mg once daily
  Other Names: Enablex
  Arms: 1
Drug: Tolterodine — Tolterodine extended release (ER) 4 mg once daily
  Arms: 2
Drug: Placebo — Placebo tablet once daily
  Arms: 3

SUMMARY:
This study will evaluate the pharmacologic effects of exposure to darifenacin and tolterodine on cardiovascular parameters in healthy subjects 50 years of age and older

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females ≥ 50 years
* Body mass index equal to or greater than 18.5 kg/m2 and less than 35.0 kg/m2

Exclusion Criteria:

* Known or suspected allergy to tolterodine ER or darifenacin or their components
* Subjects with irregular day and night patterns such as night shift workers
* Significant medical problems know to affect heart rate (ie., hypertension, hypotension, history of heart failure, history of pulmonary disease, etc.)
* History of any malignancy within the past 5 years, with the exception of localized basal cell carcinoma of the skin
* Pregnant or nursing women
* Subjects with diseases such as urinary retention, gastric retention, uncontrolled narrow-angle glaucoma, severe renal insufficiency, etc.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2006-11; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Mean heart rate per 24 hours following exposure to darifenacin 15 mg o.d. and tolterodine ER 4 mg o.d., at baseline and Day 7

SECONDARY OUTCOMES:
Effects of darifenacin and tolterodine compared to placebo on mean heart rate per 24 hours, at baseline and Day 7
Effects of darifenacin, tolterodine and placebo on other cardiovascular parameters at baseline and Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Corp., Study Chair — NPC
Locations (12):
- United States (12):
  - Investigative Site, Scottsdale, Arizona
  - Investigative Site, Tempe, Arizona
  - Investigative Site, San Diego, California
  - Investigative Site, Jacksonville, Florida
  - Investigative Site, Jupiter, Florida
  - Investigative Site, Overland Park, Kansas
  - Investigative Site, Madisonville, Kentucky
  - Investigative Site, Wellesley Hills, Massachusetts
  - Investigative Site, Hackensack, New Jersey
  - Investigative Site, Buffalo, New York
  - Investigative Site, Austin, Texas
  - Investigative Site, Dallas, Texas